CLINICAL TRIAL: NCT05416749
Title: Phase I/II Clinical Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Preliminary Antitumor Activity of 8MW2311 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Study of 8MW2311 in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor development strategy adjustment
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8MW2311-2022-CP101
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 8MW2311 (Experimental)
  Interventions: Drug: 8MW2311

INTERVENTIONS:
Drug: 8MW2311 — All subjects will receive a single intravenous (IV) infusion of 8MW2311 every 21 days (q21d), other dosing frequencies may be used.

SUMMARY:
This study is a Phase 1/2, first-in-human, open-label, dose-escalation and cohort expansion study designed to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics, preliminary antitumor activity and immunogenicity of 8MW2311 administered by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged≥18 years old;
2. Histologically or cytologically confirmed locally advanced or metastatic solid tumor;
3. Subjects must have measurable disease according to RECIST (version 1.1)；
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
5. Life expectancy >3 months;
6. Adequate organ performance based on laboratory blood tests;
7. Sexually active fertile subjects, and their partners, must agree to use methods of contraception during the study and at least 6 months after termination of study therapy；
8. Ability to understand and the willingness to sign a written informed consent document；

Exclusion Criteria:

1. History of other malignancy within 3 years before the first dose of study drug.
2. History of IL-2 or IL-2 analogues anticancer therapy.
3. Chemotherapy or radiotherapy within 21 days prior to the first dose of study drug, or any other anticancer therapy within 14 days prior to the first dose of study drug.
4. Major surgery within 28 days prior to first dose of study drug.
5. Any live vaccines within 28 days before first dose of study drug or during the study.
6. Systemic glucocorticoids or other immunosuppressants received within 14 days before first dose of study drug.
7. Toxicity related to preexisting treatment ≥Grade 2.
8. Central nervous system metastasis and/or cancerous meningitis.
9. Inadequately controlled body cavity effusions.
10. Interstitial pneumonia or interstitial lung disease, other pneumonia history or active pneumonia that may interfere with the judgement of immune-related pulmonary toxicity.
11. Active autoimmune disease, or autoimmune diseases history with recurrence possibility.
12. Clinically significant cardiac or cerebrovascular disease.
13. Use of any investigational drug within 28 days prior to the first dose of study drug.
14. Known sensitivity to any of the ingredients of the study drug.
15. Known active hepatitis B or C infection, or other serious infection.
16. History of drug abuse or drug addiction.
17. Pregnancy or lactation.
18. Other disease or condition which may put the subject at significant risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
AEs | Up to 28 days post last dose
  All the adverse events
ORR | Up to 24 months
  Objective Response Rate

SECONDARY OUTCOMES:
BOR | Up to 24 months
  Best of Response
DCR | Up to 24 months
  Disease Control Rate
CBR | Up to 24 months
  Clinical Benefit Rate
PFS | Up to 24 months
  Progression-Free Survival
DoR | Up to 24 months
  Duration of Remission
TTR | Up to 24 months
  Time to Response
TTP | Up to 24 months
  Time to Progression
OS | Up to 24 months
  Overall Survival
PK Parameter AUC | Up to 24 months
  The area under the curve (AUC)
PK Parameter Cmax | Up to 24 months
  Maximum concentration (Cmax)
PK Parameter Tmax | Up to 24 months
  Time at which maximum concentration(Tmax)
PK Parameter T1/2 | Up to 24 months
  The half life(T1/2)
Incidence of ADA | Up to 24 months
  Incidence of Anti-Drug Antibody (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - The first affiliated hospital of bengbu medicial college, Bengbu, Anhui
  - Hunan cancer hospital, Changsha, Hunan
  - Jian Zhang, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No